CLINICAL TRIAL: NCT02279914
Title: Misoprostol Dose and Timing Before Surgical Abortion at 13 to 16 Weeks' Gestation: a Randomized Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Planned Parenthood of Greater New York (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Miso
Record Dates: First submitted 2014-10-29; First posted 2014-10-31 (Estimated); Last update posted 2021-04-26 (Actual); Status verified 2021-04

CONDITIONS: Abortion, Induced
MeSH Terms: interventions — Misoprostol

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- 400 mcg (Experimental): receives 400 mcg of misoprostol 3 hours prior to the procedure
  Interventions: Drug: Misoprostol 400 mcg 3 hours prior to procedure
- 600 mcg (Experimental): receives 600 mcg of misoprostol 90 minutes prior to the procedure
  Interventions: Drug: Misoprostol 600 mcg 90 minutes prior to procedure

INTERVENTIONS:
Drug: Misoprostol 400 mcg 3 hours prior to procedure — Misoprostol 400 mcg 3 hours prior to D&E procedure
  Arms: 400 mcg
Drug: Misoprostol 600 mcg 90 minutes prior to procedure — Misoprostol 600 mcg 90 minutes prior to D&E procedure
  Arms: 600 mcg

SUMMARY:
This study is a blinded randomized trial to compare two different doses and intervals of buccal misoprostol for cervical preparation before surgical abortion at 13 to 16 weeks' gestation: 400 mcg administered 3 hours before D&E (dilation and extraction), and 600 mcg administered 1.5 hours before D&E.

Primary objective: To compare operative times after two different doses and intervals of misoprostol using a non-inferiority design.

Secondary objectives: To compare the doses and intervals of misoprostol for differences in: (1) initial cervical dilation; (2) need for mechanical dilation and ease of dilation if required; (3) ability to complete the abortion procedure without further cervical preparation; (4) complications; (5) provider variables including ease of procedure and satisfaction with cervical preparation; (6) patient variables including pre-operative side effects, post-operative pain, and acceptability

DETAILED DESCRIPTION:
The investigators compared two doses and intervals of buccal misoprostol for cervical preparation before surgical abortion at 13 to 16 weeks' gestation. This blinded randomized trial compared 400 mcg misoprostol administered 3 hours and 600 mcg administered 1.5 hours before abortion. The investigators analyzed results for the primary outcome (procedure time) using a non-inferiority limit of 3 or more minutes. The investigators tested two separate non-inferiority hypotheses each powered at 95% (2.5% confidence interval) for two gestational age groups: 13.0-14.3 and 14.4-15.6 weeks. Assuming 10% withdrawals, the investigators required 118 participants. Secondary outcomes included mechanical dilation, complications, provider satisfaction, and patient side effects and acceptability.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older
* Eligible for pregnancy termination at Planned Parenthood of NYC
* Able to give informed consent
* English speaking

Exclusion Criteria:

* Reports active bleeding, severe pain, or symptoms of spontaneous labor at enrollment
* Intrauterine fetal demise identified on pre-operative ultrasound
* Allergy to misoprostol

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2014-11; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
procedure time | day of abortion procedure
  Operative time defined as time from speculum in vagina to speculum out of vagina.

CONTACTS AND LOCATIONS:
Overall Officials: Gillian Dean, MD, MPH, Principal Investigator — Planned Parenthood of NYC
Locations (1):
- Planned Parenthood of New York City - Margaret Sanger Center, New York, New York, United States